CLINICAL TRIAL: NCT05365347
Title: Piloting of an Intervention to Reduce Problematic Alcohol Use in Early Phase Psychosis
Brief Title: Piloting of an Intervention to Reduce Problematic Alcohol Use in Early Phase Psychosis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46877
Record Dates: First submitted 2022-04-27; First posted 2022-05-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-02

CONDITIONS: Psychosis; Alcohol Use Disorder
Keywords: Early Phase Psychosis; Alcohol Use Disorder; Cognitive Enhancement Therapy
MeSH Terms: conditions — Psychotic Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: 24 participants who will be randomized to either treatment as usual in an Early Intervention for Psychosis Service (EIS) with 1 hour of psychoeducation or EIS plus cognitive enhancement therapy for alcohol misuse.
Who Masked: Outcomes Assessor
Masking Description: The psychometrist assessing participant outcomes will not be aware of the participants allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention)
- Cognitive enhancement therapy (CET) (Experimental): Cognitive enhancement therapy with an aim to reduce alcohol consumption
  Interventions: Behavioral: Cognitive Enhancement Therapy (CET)

INTERVENTIONS:
Behavioral: Cognitive Enhancement Therapy (CET) — Cognitive enhancement therapy is an evidence based intervention for schizophrenia focused on improving the cognitive domains of memory, attention span and learning ability. It has shown efficacy in reducing substance use as an indirect outcome but this will be the focus of this intervention.
  Arms: Cognitive enhancement therapy (CET)

SUMMARY:
A focus of research for youth and Emerging Adults with early phase psychosis (EPP) has been cannabis use. However, this focus has led to overlooking the possible negative influence of another legal recreational drug, alcohol. Previous studies our research group has done have demonstrated that over use of alcohol reduces the effectiveness of early intervention in psychosis treatment services. These treatment services are wrap around services that address medical, and social needs of young people with psychosis. Individuals with alcohol use disorder and EPP have fewer positive symptoms such as hallucinations which are the aspects of psychotic disorders that respond most readily to medication but have greater levels of depressive symptoms. Biologically, we can see the negative impact of alcohol on brain structure in our MRI studies. Our aim presented in this grant is to pilot a psychosocial intervention using cognitive enhancement therapy to reduce alcohol consumption in individuals with early phase psychosis. This intervention has shown promise in reducing alcohol use in individuals with long standing schizophrenia and compare it to treatment as usual which involves brief (1 session) psychoeducation. The investigators hope to reduce substance use in young people in the early stages of a psychotic disorder and improve their odds of a full recovery. In addition to measuring symptoms and hospitalizations, this trial will measure what are called social determinants of health such as return to school or work and resumption of relationships. These variables have not been measured previously in alcohol use interventions in this population but in our experience are the best indicators of long term recovery from psychosis. The symptoms will generally improve with antipsychotic drug treatment but reach a threshold after 6 months in most individuals who engage with our 5 year program. Further functional and social recovery seem to be the best determinants of a full return to health in this population.

DETAILED DESCRIPTION:
Our aim is to pilot cognitive enhancement therapy (CET) in EPP individuals with problematic alcohol use, randomizing subjects to either CET or treatment as usual (TAU), which involves brief (1 session) psychoeducation on the impacts of substance use in general on recovery. In addition to examining the impact on clinical metrics, the investigators plan to measure social determinants of health such as return to school or work and resumption of relationships. These variables have not been a focus previously in alcohol use interventions for this population, but in our experience, these measures are the best indicators of long-term functional recovery from psychosis.

This study will collect three different types of variables- demographic (things that describe the participants), clinical (things that describe how ill the individuals are) and substance use (things that measure how much or how reliant participants are on recreational substances).

Demographic variables: Age, sex, gender, ethnicity, highest education level attained and current employment or education status as well as religious status (observing/not observing/do not identify) will be collected at baseline. Employment and school enrollment will be measured again at the end of the intervention.

Clinical variables: Diagnosis will be recorded two ways, first by what the participant's clinician has determined and second for standardization, a Structured Clinical Interview from the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) will be used to give a diagnosis. Several scales will be collected, some of these are collected as part of the patient's standard of care such as the Positive and Negative Syndrome Scale (PANSS) which assesses negative and positive psychotic symptom severity, and the General Assessment of Functioning (GAF) scale which provides a broad measure of patient functioning in the domains of occupational, social and psychological functioning. These measures are collected at multiple time points in the early intervention service for psychosis.

Study specific measures are the World Health Organization Disability Assessment Schedule 2 (WHODAS 2.0), and the Psychological General Well-Being Index (PGWB) will be administered to measure by self-report the domains of anxiety, depression, general health, positive wellbeing, self-control, and vitality, measuring the impact of mental health on well-being.

Current medications will be recorded as there is some debate on the possible impact of some antipsychotic and antidepressant medications on reducing alcohol use. Health resource utilization will include hospitalizations, number of clinical appointments with the EIS and emergency room visits for the trial period. All of which can be obtained from the patient's clinician.

Substance use variables: These measures are all study specific for the timing of the collection. Hazardous alcohol use will be assessed using the World Health Organization Alcohol Use Disorders Identification Test (WHO-AUDIT) which has been used with this patient population in published studies. The WHO-AUDIT measures three areas of concern around problem drinking: amount of alcohol consumed, drinking behaviors and alcohol related problems. A total score of 8 or above is considered hazardous use. Other substance use will be measured by World Health Organization Alcohol, Smoking and Substance Involvement Screening Test (WHO-ASSIST). This measure is administered to patients when they enter the program but is not scheduled for regular use in the NSEPP. The Timeline follow-back (TLFB) will be used to collect detailed recent alcohol use over the previous 30 days history and because of its calendar approach has been shown to be very reliable in helping participants recall previous alcohol use even in individuals with a psychotic disorder. All clinical and substance use scales have been used by this research team in EPP in previous studies.

Neuropsychological profile: Cognitive enhancement therapy as the name implies was designed to help improve cognition in individuals with schizophrenia who can have problems on a number of cognitive domains which can impair functional recovery (return to school, work and relationships). Prior to the start of CET therapy, a profile of neurocognitive and psychological strengths and weaknesses must be made for each participant so that the work of the group, and homework in particular, can be targeted at domains most in need of strengthening. The neuropsychological testing will also be done on the TAU group to be able to compare the baseline values for the two groups.

Two neuropsychological composite measures will be derived from standard tests on which patients will be assessed for the best cognitive enhancement therapy modules to be used.

1. Processing speed will be quantified by measures of visual scanning ability and on reaction time. The research team will group tests from the CogState Battery for Schizophrenia (CogState Limited, New Haven, CT) which allows for measurement of these three metrics (visual scanning, simple reaction time and choice reaction time).
2. The neurocognition composite index includes measures from a variety of neurocognitive tests. The Wechsler Memory Scale which is designed to assess domains of short-term, long-term (declarative), and working memory. California Verbal Learning Test 3rd edition which as the name implies measures verbal learning and memory levels in youth and adults. The Wechsler Adult Intelligence Scale-IV to measure current intelligence quotient (IQ) scores and the National Adult Reading Test-Revised (NART-R) to give an estimate of IQ prior to illness onset. Trail making test part B with a as a measure of higher level decision making. Finally, the Wisconsin Card Sorting Test will be used to measure flexibility, and attention. Neuropsychological tests will be administered by a research assistant who is a foreign trained psychiatrist, who will be uninvolved in treatment and blinded to the treatment group of the participant.

The intervention: Individuals who consent to participate in the study will be randomized by computer algorithm to either treatment as usual (TAU) (psychoeducation) or the six month course of cognitive enhancement therapy. Randomization will be completed on a simple, secure, web-based platform (www.project-redcap.org) maintained by Nova Scotia Health (NSH) and accessible by desktop or laptop with internet access. The intervention will be bi-weekly CET sessions in a social cognitive group format over a six month period. The basis of CET is a developmental, small-group approach to improving learning and memory; as well as social intelligence (the ability to gauge others' social reactions for instance) and this has been shown to reduce alcohol use in individuals with longer standing schizophrenia. The therapy is manualized and has recognition from Substance Abuse and Mental Health Services Administration (SAMHSA) in the USA as an effective therapy in individuals with schizophrenia for overall learning and memory improvement. Homework and psychoeducation are a feature of this therapy. Therefore, the investigators have chosen a brief psychoeducation alone intervention in addition to TAU in an early intervention service as the treatment control for this study. The control group will have a one hour psychoeducation session based on the impact of alcohol use on the brain and on recovery in individuals with a psychotic disorder. The length of this therapy is less than the approach in individuals with chronic schizophrenia who have a more significant illness burden, and with the aim of reducing attrition from the therapy; hence our labeling of this as a pilot study both for the population under study and re-working of the intervention into a time window that has been shown to work more effectively for patient engagement.

The trial is planned as follows: one set of 12 CET and 12 TAU participants will start the trial then two months later a second set of 12 CET and 12 TAU will begin the trial. Enrollment of 12 individuals per group should account for our estimated dropout rate for this shortened delivery of between 30-40%. This approach should ensure completion of the trial by 8 individuals per group. Participant attendance at each session will be recorded as well as measure of engagement to the therapy such as completion of homework.

Treatment as Usual group: Enrollment in an early intervention service (EIS) has been shown to reduce substance use up to 25% for cannabis use but it is not well studied if alcohol use is similarly reduced. EIS offer intensive supportive care and psychoeducation for substance use so this will be our control group

ELIGIBILITY:
Inclusion Criteria:

* This study will enroll individuals 16-35 years of age from Early Intervention Services for Psychosis in Nova Scotia
* less than 5 years of psychotic illness.
* Individuals will have a psychotic spectrum diagnosis (primary psychotic disorder) that will include schizophrenia, schizoaffective disorder, and unspecified schizophrenia spectrum disorder.
* have problematic alcohol use (score of 8 or higher on the World Health Organization Alcohol Use Disorders Identification Test (WHO-AUDIT))

Exclusion Criteria:

* presence of another substance use disorder other than nicotine dependence

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption (mL per day) | 6 months
  To determine if youth and emerging adults with early phase psychosis and problematic alcohol use (score of 8 or higher on the AUDIT) will reduce alcohol consumption after treatment with a cognitive enhancement therapy intervention. Changes in alcohol consumption will be measured (mL per day).

SECONDARY OUTCOMES:
Feasibility of a shortened intervention | 6 months
  To measure the feasibility of a modified CET approach in an early psychosis patient population by measuring patient engagement and trial retention. The number of sessions completed by each participant will be recorded (attendance in weeks).
Possible role of gender in alcohol consumption | 6 months
  To measure whether women benefit equally from cognitive enhancement therapy compared to men. Changes in the level of alcohol used from start to end of trial (measured in mL per day) will be compared across gender groups to see if there are differences in therapeutic response to this intervention between men and women.
Engagement based on gender | 6 months
  To examine the level of engagement or comfort that men and women have with the intervention, we will measure the level of attendance for CET sessions by men and women enrolled in the trial. The percentage completing the trial in both gender groups will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Tibbo, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The ability to share IPD is currently undecided as it will be based on the decision of the privacy office at our institution. This protocol will be updated after review.